CLINICAL TRIAL: NCT03170180
Title: Exploratory Study of Drug Sensitivity Prediction Software (IRCR-DReSS) With Patient-derived Tumor Cells of Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-12-058
Record Dates: First submitted 2017-05-26; First posted 2017-05-30 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Sunitinib; Gefitinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sunitinib (Experimental)
  Interventions: Drug: Sunitinib
- gefitinib (Experimental)
  Interventions: Drug: Gefitinib
- imatinib (Experimental)
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Sunitinib — sunitinib 37.5mg daily
  Arms: sunitinib
Drug: Gefitinib — Gefitinib 250mg daily
  Arms: gefitinib
Drug: Imatinib — Imatinib 400mg daily
  Arms: imatinib

SUMMARY:
1. Metastatic gastric cancer patients who failed standard treatment will be enrolled in this study.
2. After consent form, patient-derived cancer cell will be collected and tested with 3 kinds of drugs (sunitinib, gefitinib, imatinib).
3. Drug sensitivity prediction software (IRCR-DReSS) will present level of sensitivity and patients will be treated with sensitive drugs.
4. Patients will be evaluated every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age>-20
* metastatic gastric cancer
* life expectancy >-3 months
* ascites and pleural effusion that can be drained
* ECOG 0-2
* Proper organ function
* Patients who will be enrolled in sunitinib, gefitinib, imatinib clinical trial

Exclusion Criteria:

* HBeAg, HCV, HIV (+)
* Active infection
* Uncontrolled systemic disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided